CLINICAL TRIAL: NCT03002467
Title: Impact Analysis of Prognostic Stratification for Pulmonary Embolism: A Randomized Controlled Trial
Brief Title: Impact Analysis of Prognostic Stratification for Pulmonary Embolism
Acronym: iAPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Alessandro Squizzato, Associate Professor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: iAPP study
Record Dates: First submitted 2016-12-11; First posted 2016-12-23 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

ARMS (2):
- PESI score (Experimental): treating physicians must formally calculate PESI and report in the clinical record form* each day of hospitalization on top of routine clinical practice (standard care)
  Interventions: Other: PESI score
- Standard care (No Intervention): standard care (i.e. no formally calculation of PESI on top)

INTERVENTIONS:
Other: PESI score
  Arms: PESI score

SUMMARY:
The Investigator postulate that the use of PESI in addition to routine clinical practice, as opposed to routine clinical practice based on clinical judgment alone, will help physicians to correctly identify PE patients at low-risk of adverse outcomes. Considered that low-risk patients could benefit from a short hospital stay, aim of this study is to demonstrate that the use of PESI will lead physicians to discharge these patients earlier, thus reducing the duration of hospital stay of PE patients (primary outcome).

Outpatients diagnosed with PE at the emergency department (ED) and admitted to participating units represent the target population

As the availability of DOACs may influence the duration of hospital stay, the secondary objectives of the present study are:

1. to demonstrate that a shorter hospital stay for low-risk PE patients (independently on the method used to identify them) will reduce the incidence of hospital-associated complications and improve patients satisfaction and quality of life, without increasing the incidence of PE-related complications
2. to demonstrate that the use of PESI, as opposed to clinical judgment alone, will be associated with a greater proportion of patients discharged early (< 72 hours from ED admission) or treated entirely at home (< 24 hours from ED admission).
3. to demonstrate that the use of DOACs will reduce the duration of hospital stay of PE patients
4. to demonstrate that the use of DOACs, as opposed to standard treatment, will be associated with a greater proportion of patients discharged early (< 72 hours from ED admission) or treated entirely at home (< 24 hours from ED admission).

DETAILED DESCRIPTION:
STUDY DESIGN

Within 24 hours from acute PE diagnosis, each treating physician (local Investigator) will be centrally randomized. Treating physicians (local Investigator) of the participating Units will call the coordinating centres by phone for randomization. Before randomization, in order to avoid any influence on treatment choice, each treating physician (local Investigator) should declare in advance which treatment strategy will use for his patient (intention-to-treat), i.e. standard treatment with heparin plus vitamin K antagonist (standard group) or DOACs (DOACs group) Randomization will be stratified by treatment choice of the local Investigator. Each of two 'intention-to-treat' approaches will be therefore randomized to two arms, i.e. arm 1 or arm 2.

Arm 1: treating physicians must formally calculate PESI and report in the clinical record form* each day of hospitalization on top of routine clinical practice (standard care)

Arm 2: standard care (i.e. no formally calculation of PESI on top)

Randomization will be performed centrally with a 1:1 ratio, following a computer-generated list of randomization.

STUDY POPULATION

1.1 Population

Randomised physicians:

Each Local Investigator of participating canters. All participating centres are Internal Medicine Unit.

PE population:

Consecutive adult outpatients of any age, gender and race, with an objectively confirmed diagnosis of a suspected or unsuspected acute PE at the emergency department (ED) and admitted to participating units will be included.

Suspected PE means that diagnosis has been made by an imaging test (computed tomographic pulmonary angiography [CTPA], pulmonary angiography, V/Q lung scan) prescribed by a treating physician who had clinical suspicion of PE.

Unsuspected PE means that diagnosis has been made incidentally by an imaging test performed for other clinical indications (e.g. cancer staging or follow-up).

Objective diagnosis of acute PE means: a positive computed tomographic pulmonary angiography (CTPA), a positive pulmonary angiography, a high-probability V/Q lung scan (or perfusion lung scan with negative chest X-ray), or intermediate probability V/Q or perfusion lung scan with proximal deep-vein thrombosis (DVT) documented by compression ultrasonography.

1.2 Sample size calculation

The Investigators hypothesize that the distribution of hospital stay duration for PE will have a standard deviation of 4 days. The I vestigators also hypothesize that the mean duration of hospital stay will be reduced by at least 15% in PE patients whose treating physician will be randomised to formally use PESI and by 5% in PE patients whose treating physician will not be randomised to formally calculate PESI. Low-risk PE patients are almost 50% of all PE population. Therefore, with an α error of 0.05 and a statistical power (1-β error) of 80%, 200 patients for each group (a total of 400 patients) need to be enrolled to find a statistically significant difference (p<0.05) between the mean hospital stay length. As the variable 'hospital stay length' will have a non-normal distribution and needs to be expressed and reported as median, 10% extra patients need to be enrolled to reach a statistically significant difference with the previous statistical assumptions.

Final total sample size will be, therefore, of 440 patients (220 patients for each group)

OUTCOMES

1. Main study parameter/endpoint

   The primary outcome is the median length of hospital stay
2. Secondary study parameters/endpoints

The secondary efficacy outcomes will be the following:

1. health-system measures

   * proportion of patients undergoing short-hospital stay
   * proportion of patients undergoing complete home-treatment
   * post-discharge hospital re-admission
   * post-discharge outpatient visits to emergency department
2. patient-related outcomes

   * quality of life (5-point Likert scale questionnaire)

The safety outcomes will be the following:

1. overall mortality
2. PE-related

   * PE-related mortality
   * recurrent PE and/or deep vein thrombosis (DVT)
   * major bleeding
   * clinically relevant non-major bleeding
   * minor bleeding
   * other anticoagulation-related complications (hematoma/infection at heparin or fondaparinux injection sites, heparin-induced thrombocytopenia)
3. Hospitalization-related

   * hospital-acquired infections (pneumonia; urinary tract infection; other)
   * iatrogenic complications
   * immobilization syndrome
   * pressure sores

Overall mortality, PE-related safety outcomes, post-discharge hospital re-admission and outpatient visits to emergency department will be measured at 14 days, 30 days, and 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with objectively diagnosed PE, both suspected or unsuspected (e.g. during CT for cancer staging and/or follow-up)
* Age > 18 years
* Signature of written informed consent

Exclusion Criteria:

* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Squizzato, MD PhD, Principal Investigator — Università degli Studi dell'Insubria
Locations (1):
- Cuneo, Italy

REFERENCES:
- [Derived] Donadini MP, Mumoli N, Fenu P, Pomero F, Re R, Palmiero G, Spadafora L, Mazzi V, Grittini A, Bertu L, Aujesky D, Dentali F, Ageno W, Squizzato A. The Clinical Impact of the Pulmonary Embolism Severity Index on the Length of Hospital Stay of Patients with Pulmonary Embolism: A Randomized Controlled Trial. Diagnostics (Basel). 2024 Apr 7;14(7):776. doi: 10.3390/diagnostics14070776. PMID 38611689